CLINICAL TRIAL: NCT03664622
Title: Does Low-Dose Ketamine Infusion or Intravenous Morphine Infusion During Abdominoplasty Change Postoperative Pain Profile? : A Double-Blind, Randomized, Controlled Clinical Trial
Brief Title: Ketamine Versus Morphine Change Pain Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hassan Mohamed Ali, associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: wahdan kteamine
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Ketamine; Morphine

STUDY DESIGN:
Intervention Model Description: ketamine versus morphine
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group K (Experimental): patients with a ketamine infusion intraoperative
  Interventions: Drug: Ketamine
- group M (Experimental): patients with a Morphine infusion intraoperative
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Ketamine — Ketamine group to whom intravenous ketamine was administered in a loading dose of 0.15 mg/kg over 5 min, 10 minutes pre incision, followed-by an infusion at 2 micg/kg/min until the end of surgery.
  Other Names: Ketamine infusion
  Arms: group K
Drug: Morphine — a loading dose of 0.1 mg/kg over 20 min intravenously, 10 minutes pre incision, then infused with morphine an infusion rate of 5 - 40 microgram/kg/hour till the end of surgery.
  Other Names: Morphine infusion
  Arms: group M

SUMMARY:
The aim of this study is to evaluate the efficacy of intravenous low dose ketamine infusion versus morphine infusion analgesia for pain reduction in Abdominoplasty surgery

DETAILED DESCRIPTION:
Abdominoplasty is considered one of the most commonly performed cosmetic procedures. According to statistics from the International Society of Aesthetic Plastic Surgery, a total of 758,590 abdominoplasties were performed in the world in 2016. This is an increase of 72.95% in comparison with 2011, making it the fourth most common cosmetic procedure. Given the increasing number of abdominoplasties performed, the importance of understanding the possible complications and morbidity associated with the procedure is critical. One of these complications is the postoperative pain. With adequate postoperative pain control, the patients met discharge criteria sooner and this helps in shortening the hospital stay, better overall patient satisfaction, and decreased hospital costs. Therefore, the severity of this problem and the all drug agent used to prevent and treat postoperative pain best interest to be aware in the anesthesiologists. Traditionally, analgesia for abdominal wall surgery is provided either by systemic drugs such as opioids, nonsteroidal anti-inflammatories, alpha 2 agonists and paracetamol or by epidural analgesia. However, Opioids, such as morphine or fentanyl, remain the mainstay of postoperative analgesic regimens for patients after abdominal wall surgery. The pain is not always fully relieved by such agents, and often patients develop tolerance to them. The ever-increasing doses of opioids are clearly not without their adverse effects. (5) For this Alternative approaches, which reduce the requirement for strong opioids post-operative, are required. Recently, interest has focused on the use of N-methyl-D-aspartate (NMDA) receptor antagonists for the management of postoperative pain. Ketamine exerts its main analgesic effect by antagonism of NMDA receptors that not only abolishes peripheral afferent noxious stimulation, but it may also prevent central sensitization of nociceptors as shown in animal studies with the excellent analgesic property even in subanesthetic doses. (6) Various recently published studies have talked about the analgesic effect of low-dose ketamine (7,8) however, all of this study are relatively short procedure time, reduced surgical stimulation and small sample size. The aim of this study is to evaluate the efficacy of intravenous low dose ketamine infusion versus morphine infusion analgesia for pain reduction in Abdominoplasty surgery

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II
* patients aged between 18-50 years old. -

Exclusion Criteria:

* those who refused to participate
* ASA physical status III, IV, patients younger than 18 years or older than 50 years old
* super morbid obesity with BMI 50, history of epilepsy
* patients having a history of parenteral or oral analgesics within the last 24 hours before
* initiation of operation
* those having an allergy to study agents.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
dose of fentanyl | 4 hours
  Amount of fentanyl needed intraoperative and postoperative after extubation, and every hour postoperative for four hours.

SECONDARY OUTCOMES:
pain assessment: VAS (Visual analogue scale) | 4 hours
  Visual analogue scale for pain assessment.( VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom,pain,health) orientated from the left (worst) to the right (best). In some studies,horizontal scales are orientated from right to left ,and many investigators use vertical VAS.The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom,pain,health) orientated from the left (worst) to the right (best). In some studies,horizontal scales are orientated from right to left .

OTHER OUTCOMES:
patient sedation (Ramsey Scale for assessment of patient sedation) | 4 hours
  Anxious agitated and restless= 1 point
  * Cooperative, oriented and tranquil= 2 points
  * Responding only to verbal commands= 3 points
  * Brisk response to light glabella tap or loud auditory stimulus= 4points
  * Sluggish response to light glabella tap or loud auditory response= 5 points
  * No response to light glabella tap or loud auditory response= 6 points

CONTACTS AND LOCATIONS:
Overall Officials: hassan Ali, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No